CLINICAL TRIAL: NCT06074679
Title: Clinical Study of Single Incision Laparoscopic Cholecystectomy in the Treatment of Patients With Acute Cholecystitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Changxing Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University (Unknown); Suichang Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University (Unknown); Jiande Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University (Unknown); Shexian Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-0690
Record Dates: First submitted 2023-09-23; First posted 2023-10-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: Single-incision laparoscopic cholecystectomy; Conventional laparoscopic cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-incision laparoscopic cholecystectomy (Experimental): SILC was defined as laparoscopic surgery done through a single trans-umbilical incision
  Interventions: Procedure: Open cholecystectomy
- Conventional laparoscopic cholecystectomy (Active Comparator): CLC was defined as three or four port surgery carried out with either French or American position.
  Interventions: Procedure: Open cholecystectomy

INTERVENTIONS:
Procedure: Open cholecystectomy — The experimental group and the control group were changed to open cholecystectomy when the operation was difficult to complete.

SUMMARY:
Gallstone is a common disease in China.At present, the prevalence of gallstones in China is 15 %, and about 210 million people are sick. Acute cholecystitis is acute gallbladder inflammation, is one of the main complications of cholelithiasis or gallstones. The removal of gallbladder and gallstones in patients with acute cholecystitis in the presence of biliary pain will prevent the recurrence of gallbladder and reduce the risk of cholecystitis progression. If gallbladder perforation is not treated in time, the mortality rate is 30 %. Acute acalculous cholecystitis without treatment will be life-threatening, with a mortality rate of up to 50 %. At present, the vast majority of patients with acute cholecystitis are treated with 4-hole traditional laparoscopic cholecystectomy and open cholecystectomy. Their postoperative quality of life, pain and scar-related complications, remain major factors for patients.In recent years, with the renewal of the concept of minimally invasive surgery and the continuous advancement of instruments and technology, single-incision laparoscopic cholecystectomy has also maximized the quality of life after surgery and reduced postoperative pain and scar-related complications. At present, there are few reports on randomized controlled clinical trials of SILC in patients with acute cholecystitis, and there is a lack of large sample size studies.Due to the difficulty of SILC operation, the longer learning curve, the different equipment conditions and technical characteristics of each center, and the lack of standardized training, there is no effective consensus on the application indications and operation procedures of SILC in acute cholecystitis surgery. Based on the current status, the purpose of this study was to investigate the effect of SILC on postoperative quality of life, postoperative pain, scar assessment and postoperative complications in patients with acute cholecystitis, so as to propose a standardized single incision laparoscopic operation procedure in the treatment of acute cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* Acute cholecystitis（GradeⅠ，II）

Exclusion Criteria:

* Combined with liver cirrhosis (Child grade B and above)
* Upper abdominal surgical history;
* Changes in surgical plan (conversion to laparotomy,cholangiography, bile duct exploration, bile duct injury repair, abscess clearance, multivisceral resection.)
* Patients and their families do not agree with the treatment lost follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (time to return to normal life) | 3 years
  The quality of life of patients after operation was investigated by a unified SF-36 questionnaire. The higher the final score, the better the quality of life.

SECONDARY OUTCOMES:
Cosmetic result | 3 years
  Evaluation of postoperative incisional scarring using the Vancouver Scar Scale. The lower the score, the higher the scar satisfaction.

OTHER OUTCOMES:
Grade II or above incidence of complications | 3 years
  Postoperative complications were defined by the clavien-dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Daren, MD, PhD, Study Director — Chief Physician
Locations (5):
- China (5):
  - Shexian Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University, Huangshan City, Anhui
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang
  - Changxing Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University, Huzhou, Zhejiang
  - Suichang Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University, Lishui, Zhejiang
  - Jiande Branch, Second Affiliated Hospital, School of Medicine, Zhejiang University, Meicheng, Zhejiang

IPD SHARING:
Plan to Share IPD: No